CLINICAL TRIAL: NCT02328573
Title: The Impact of Group Singing on Patients With Stroke and Their Personal Caregivers
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Joanne Loewy, Associate Clinical Professor, Family Medicine & Community Health, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-1215; 001-14 (Other: Beth Israel Medical Center)
Record Dates: First submitted 2014-06-23; First posted 2014-12-31 (Estimated); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Stroke and Aphasia
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Communal singing (Experimental): Participants in the study group will join the choir and participate in a weekly hour rehearsal for six months and will be assessed for aphasia, mood, and quality of life outcomes
  Interventions: Behavioral: Communal singing
- Control (No Intervention): The control group will not participate in the choir for the first six months. At the end of the six months study period, all participants will be evaluated again for changes in aphasia, language, mood and quality of life

INTERVENTIONS:
Behavioral: Communal singing
  Arms: Communal singing

SUMMARY:
The study will focus on the impact of communal singing on patients with stroke and their personal caregivers. Forty post-stroke patients will be randomly assigned to two groups: the first group of 20 stroke survivors and their caregivers (up to 40 total participants) will receive 6 months (approximately 24 sessions) of music therapy. The second control groups of 20 stroke survivors and their caregivers will receive standard post-stroke care

DETAILED DESCRIPTION:
The study will focus on the impact of communal singing on patients with stroke and their personal caregivers. Forty post-stroke patients will be randomly assigned to two groups: the first group of 20 stroke survivors and their caregivers (up to 40 total participants) will receive 6 months (approximately 24 sessions) of music therapy. The second control groups of 20 stroke survivors and their caregivers will receive standard post-stroke care.

All enrolled participants will be assessed on their mood, past music experience and music genre preference (music therapy assessment). They will complete the abridged Beck (BDI-2-fastscreen) questionnaire, the stoke and aphasia quality of life scale; a Likert which measures distress; the Western Aphasia Battery (WAB); the NIH Stroke Scale (SS); the Figely compassion scale; and the driving scene test (Stern and White); and the Rankin. In additional we will take saliva samples from all participants to measure hormone levels.

Participants can attend zoom or live.

ELIGIBILITY:
Inclusion Criteria:

* Stroke victim, regardless of level of stroke

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-04-04 (Actual); Primary Completion 2025-06-09 (Actual); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Change in mood and quality of life as indicated through saliva (cortisol and melatonin sampling) | 6 months
  Cortisol and melatonin sampling will be conducted at baseline and at 6 months

SECONDARY OUTCOMES:
Change in language aphasia outcome improvement | 6 months
  We will use the following scales as 6 month measurements, and will compare these scores to the initial assessments: Speech Therapy Evaluation-Western Aphasia Battery NIH Stroke Scale and Aphasia Quality of Life Scale.

OTHER OUTCOMES:
Change in motivation and verbal expression | 6
  We will use the following scales as 6 month measurements, and will compare these scores to the initial assessments: Likert Scale Mood (Beck-BDI 2)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Loewy, DA, Principal Investigator — Beth Israel Medical Center
Locations (1):
- Mount Sinai Beth Israel, New York, New York, United States